CLINICAL TRIAL: NCT02938260
Title: Diltiazem vs. Metoprolol in the Acute Management of Atrial Fibrillation in Patients With Heart Failure With Reduced Ejection Fraction
Brief Title: Diltiazem vs. Metoprolol in the Acute Management of AF in Patients With HFrEF
Status: Completed | Type: Observational
Sponsor: RaeAnn Hirschy (Other)
Responsible Party: Sponsor-Investigator, RaeAnn Hirschy, PGY2-Critical Care, Rush University Medical Center
Organization: Rush University Medical Center (Other)
Other Study IDs: 16090607
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Atrial Fibrillation; Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Diltiazem
  Interventions: Drug: Metoprolol vs Diltiazem
- Metoprolol
  Interventions: Drug: Metoprolol vs Diltiazem

INTERVENTIONS:
Drug: Metoprolol vs Diltiazem

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia, accounting for one third of all hospital admissions and 1% of all emergency department visits (ED). Approximately 65% of those presenting to the ED with AF are admitted. There are also numerous reasons for patients to get AF with rapid ventricular rate (AF RVR) during hospitalization. In the acute setting these patients are often treated with diltiazem, a non-dihydropyridine calcium channel blocker (ND CCB), or metoprolol, a beta blocker (BB). Non-dihydropyridine calcium channel blocker (diltiazem and verapamil) use is considered harmful and national guidelines recommend against use in patients with decompensated heart failure (HF). This recommendation is based on studies with long-term treatment. The purpose of this study is to assess the difference between metoprolol and diltiazem for the acute treatment of AF RVR in patients with HF with reduced ejection fraction (HFrEF).

DETAILED DESCRIPTION:
AF and HF are frequently seen in the hospital setting. AF affects over 2 million people in the United States, while HF affects over 5 million. These disease states have a significant morbidity and mortality impact with AF leading to a 4 fold increase in stroke and 2 fold increase in death, while 50% of patients with a new HF diagnosis will die within 5 years. These two disease states share several common risk factors including, age, hypertension, diabetes mellitus, and heart disease. Based on this relationship and the changes in myocardial structure, function, and conduction the two are also risk factors for one another. Of patients with HF, 61.5% of men and 73% of women develop AF. Of those with AF, 73% of men and 75.6% of women develop HF.

Both the AF guidelines by the American Heart Association, American College of Cardiology, and Heart Rhythm Society and the HF guidelines by the American College of Cardiology Foundation and the American Heart Association recommend against the use of ND CCB in patients with HFrEF. The HF guidelines specify to avoid ND CCB in patients with reduced LVEF, but also mention avoiding most calcium channel blockers in general with the possible exception of amlodipine, due to known adverse effects and potential for harm. However, short term use of diltiazem for the acute control of RVR in patients with HFrEF has not been clearly evaluated. Three studies compare the use of BB and ND CCB in the acute treatment of AF RVR. These studies excluded those with severe (New York Heart Association Class IV) or decompensated HF, however, they did not comment on patients with compensated HFrEF. Most of these studies illustrate no difference, but the most recent study reported a success rate (heart rate (HR) <100 bpm within 30 minutes) of 95.8% with intravenous (IV) diltiazem and 46.4% with IV metoprolol (p<0.0001).

When comparing use of long term and short term therapy in patients with HFrEF a different perspective emerges. Both BB and ND CCB have negative inotropic effects which can be harmful during an acute HF exacerbation and worsen symptoms. However, BB are routinely recommended for chronic use in HFrEF due to their added neurohormonal benefit, which over time delays HF progression and reduces mortality. In contrast, long term treatment with ND CCB in those with pulmonary congestion is associated with an increased cumulative rate of cardiac events (hazard ratio 1.41). The comparative short term benefit in patients is still unclear. In a small study, patients with AF RVR and severe HF, 97% treated with IV diltiazem had a HR reduction of >20% and no evidence of HF exacerbation. A second study of patients in decompensated HF compared the use of IV metoprolol and diltiazem for control of AF RVR. Both agents were equally effective at controlling heart rate with no difference in safety endpoint or evidence of worsening heart failure. Neither of these studies specifically address compensated HFrEF.

Current literature focuses on the risks associated with ND CCB and patients with HFrEF, but these effects are with long-term treatment. Studies in the acute setting often exclude those with severe or decompensated HFrEF. Therefore, a study focusing on metoprolol versus diltiazem for the acute control of AF RVR in patients with HFrEF could offer an insight into current clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant adults ≥18 years of age with AF RVR (HR >120 bpm), which will be obtained from vital signs or electrocardiogram, in the emergency department, who have an EF <40% from an echocardiogram within the previous 4 years, and are treated with IV push metoprolol or diltiazem as first line for rate control of AF with RVR. Patients can receive up to two IV push doses but cannot switch treatment medication between these two doses.

Exclusion Criteria:

* Patients with a SBP <90 mmHg or decompensated heart failure (ie those presenting primarily with worsening of heart failure signs and symptoms, including dyspnea and lower extremity edema). Patients who are admitted multiple times within the time frame or have multiple episodes will be excluded except for the first episode within the first admission.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: To compare the achievement of a goal heart rate of <100 bpm or a HR reduction of at least 20% in patients with HFrEF receiving intravenous diltiazem versus intravenous metoprolol for rate control of AF with RVR.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Successful rate control | 30 minutes
  Successful rate control within 30 minutes from the first dose (HR <100 bpm or a decrease by at least 20%).

SECONDARY OUTCOMES:
Successful rate control within 15 minutes | 15 minutes
  Successful rate control within 15 minutes
Successful rate control within 60 minutes | 60 minutes
  Successful rate control within 60 minutes
Bradycardia | 30 minutes
  HR <60 bpm
Hypotension | 30 minutes
  SBP <90 mmHg
Conversion | 30 minutes
  conversion to sinus rhythm
Worsening heart failure symptoms | 48hr/readmission
  new inotropic support, new pulmonary edema, or increased O2 requirement within 48 hr or readmission within 7 days of discharge